CLINICAL TRIAL: NCT02736513
Title: Pilot, Phase 2 Study Assessing Intracranial Activity of AZD9291 (TAGRISSO) in Advanced EGFRm(EGFR Mutation) NSCLC Patients With Asymptomatic Brain Metastases
Brief Title: Intracranial Activity of AZD9291 (TAGRISSO) in Advanced EGFRm NSCLC Patients With Asymptomatic Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Nir Peled MD, PhD, Head of Oncology, Shaare Zedek Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-15-11084
Record Dates: First submitted 2016-03-22; First posted 2016-04-13 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Lung Cancer
Keywords: Tagrisso; AZD9291; EGFRm; brain metastases; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD9291 80 mg - naive patients (Experimental): naive patients with tumors harbouring either exon 19 deletion, L858R, T790M, or uncommon sensitizing EGFR mutations, will be treated with AZD9291 80 mg/day
  Interventions: Drug: AZD9291
- AZD9291 80 mg - previously treated T790M was diagnosed (Experimental): Patients previously treated with first and second generation EFGR TKIs (either Gefitinib, Erlotinib or Afatinib) in whom T790Mwas diagnosed either in the tumor specimen or in the ctDNA after testing it following the most recent disease progression, will be treated with AZD9291 80 mg/day
  Interventions: Drug: AZD9291
- AZD9291 80 mg - previously treated unrelated to T790M (Experimental): patients advanced NSCLC previously treated with 1st/2nd generation EGFR TKIs (either gefitinib. erlotinib or afatinib) who progressed unrelated to T790M (T790M-). No restriction regarding the number of prior EGFR TKIs or cytotoxic chemotherapy lines of treatment is applied.
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291 — Patients will receive AZD9291 at a dose of 80 mg once daily.
  Other Names: TAGRISSO

SUMMARY:
Patients will receive AZD9291 at a dose of 80 mg once daily. Intracranial response will be assessed with brain MRI scan, systemic evaluation will be done by PET-CT (Positron Emission Tomography-Computed Tomography) scan.

In case of isolated CNS progression which may or may not be accompanied by asymptomatic systemic progression, AZD9291 dose will be escalated to 160 mg once daily. For patients whose intracranial disease will progress further, brain radiotherapy (in the form of SRS or WBRT) will be administered; treatment with AZD9291 will be interrupted and re-initiated at a standard dose after the end of radiotherapy course in the absence of symptomatic systemic progression. The treatment will be continued until symptomatic systemic progression, unacceptable toxicity or further intracranial progression following brain radiotherapy administration (whichever occurs first). All patients will be followed until death or 5 years.

DETAILED DESCRIPTION:
Patients will receive AZD9291 at a dose of 80 mg once daily. Intracranial response will be assessed with brain MRI scan, systemic evaluation will be done by PET-CT scan. In case of isolated CNS progression which may or may not be accompanied by asymptomatic systemic progression, and having in mind the blood-brain-barrier as a possible pharmacokinetic resistance mechanism here, AZD9291 dose will be escalated to 160 mg once daily. For patients whose intracranial disease will progress further, brain radiotherapy (in the form of SRS or WBRT) will be administered; treatment with AZD9291 will be interrupted and re-initiated at a standard dose after the end of radiotherapy course in the absence of symptomatic systemic progression. The treatment will be continued until symptomatic systemic progression, unacceptable toxicity or further intracranial progression following brain radiotherapy administration (whichever occurs first). All patients will be followed until death or 5 years.

Intracranial outcomes will be assessed by modified RECIST criteria (mRECIST) and analyzed. The added value of the increased dose (160 mg) after failure of the standard dose will be assessed as well. Since only neurologically asymptomatic patients are planned to be enrolled, it is important to use mRECIST criteria which allows small brain lesions to be assessed (according to these criteria, ≥ 5mm tumors are considered measurable and up to 5 target lesions are allowed) 1. Systemic response assessment will be done using RECIST 1.1. Exploratory analysis of the outcomes will be performed according to the treatment setting ( treatment-naïve vs. acquired resistance setting) and EGFR mutation subtype. Additionally, serum protein biomarker analysis will be performed in correlation with intracranial and systemic response. Safety parameters will be monitored.

ELIGIBILITY:
1. Provision of informed consent prior to any study specific procedures
2. Male or female, aged at least 18 years.
3. Group A: treatment-naïve advanced NSCLC with an sensitizing EGFR mutation.

   * Patients who received adjuvant/neo-adjuvant chemotherapy/chest irradiation/palliative irradiation (other than brain) allowed.
   * Exon 19 deletion, L858R, T790M and uncommon sensitizing EGFR mutations in treatment-naïve patients are allowed.

   Or

   Group B: patients advanced NSCLC previously treated with 1st/2nd-generation EGFR TKIs (either gefitinib. erlotinib or afatinib) in whom T790M was diagnosed in the tumor specimen or ctDNA after testing it following the most recent disease progression.
   * No restriction regarding the number of prior EGFR TKIs or cytotoxic chemotherapy lines of treatment is applied.
   * Group C: patients advanced NSCLC previously treated with 1st/2nd generation EGFR TKIs (either gefitinib. erlotinib or afatinib) who progressed unrelated to T790M (T790M-). No restriction regarding the number of prior EGFR TKIs or cytotoxic chemotherapy lines of treatment is applied.
4. Asymptomatic untreated brain metastases (previously SRS more than 6 month).
5. Measurable intracranial disease by mRECIST criteria (less or equal to 5 mm).
6. Normal hematologic, renal and liver function:

   Absolute neutrophil count above 1500/mm3, platelets above 100,000/mm3, hemoglobin above 9 g/dL; createnine concentration is less or equal to 1.5 mg/dL, or createnine clearance less then 60 ml/min. Total bilirubin less or equal to 1.5 mg/dL, ALT+ AST levels 5 times above the upper normal limit.
7. World Health Organization (WHO) performance status 0-2.
8. Patients must have a life expectancy ≥ 12 weeks.
9. Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
11. All patients with reproductive potential must agree to use barrier contraception methods while receiving the study treatment.
12. Patients has the ability to read and write and use the electronic devices.
13. At least one lesion (measurable and/or non-measurable) that can be accurately assessed by CT/MRI at baseline and follow up visits.

3.2 Exclusion criteria

1. Involvement in the planning and/or conduct of the study (applies to both sponsor staff and/or staff at the study site).
2. Previous treatment with AZD9291.
3. Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inhibitors of CYP3A4 (at least 1 week prior) and potent inducers of CYP3A4 (at least 3 week prior) (Appendix A). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer/inhibitory effects on CYP3A4.
4. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy.
5. EGFR TKI - resistant EGFR mutations (e.g., insertion in exon 20).
6. T790M is allowed.
7. Patients previously treated with WBRT.
8. Pregnant or lactating women.
9. Inability to sign the informed consent form.
10. Any concurrent and/or other active malignancy that has required systemic treatment within 2 years of first dose of study drug.
11. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV), uncontrolled diabetes.
12. Inability to swallow the formulated product, malabsorption syndrome, refractory nausea and vomiting that would preclude adequate absorption of AZD9291.
13. Any of the following cardiac criteria:

    1. Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 consequent ECGs, using the screening clinic ECG machine-derived QTc value;
    2. Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG;
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, including unexplained sudden death under 40 years of age in a first-degree relative, or any concomitant medication known to prolong the QTc interval.
14. Any evidence/past medical history of cardiomyopathy.
15. Any evidence/past medical history of interstitial lung disease (ILD) or radiation pneumonitis which required steroid treatment.
16. History of hypersensitivity to AZD9291 (or drugs with a similar chemical structure or class to AZD9291) or any excipients of these agents
17. Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry
18. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Intracranial overall response rate as defined by modified RECIST | 5 years
  Patients will receive TAGRISSO. Intracranial response will be assessed with brain MRI scan, systemic evaluation will be done by PET-CT scan.

SECONDARY OUTCOMES:
Intracranial disease control rate (IDCR) as defined by mRECIST | 5 years
  Patients will receive TAGRISSO. Intracranial response will be assessed with brain MRI scan, systemic evaluation will be done by PET-CT scan.
median time to intracranial response (mTTIR) as defined by mRECIST | 5 years
  Patients will receive TAGRISSO. Intracranial response will be assessed with brain MRI scan, systemic evaluation will be done by PET-CT scan.
median intracranial progression free survival (mIPFS) as defined by mRECIST | 5 years
  Patients will receive TAGRISSO. Intracranial response will be assessed with brain MRI scan, systemic evaluation will be done by PET-CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Peled, MD PhD FCCP, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Peled N, Kian W, Inbar E, Goldstein IM, Zemel M, Rotem O, Rozenblum AB, Nechushtan H, Dudnik E, Levin D, Zer A, Keren-Rosenberg S, Yust-Katz S, Fuchs V, Remilah AA, Shelef I, Roisman LC. Osimertinib in advanced EGFR-mutant lung adenocarcinoma with asymptomatic brain metastases: an open-label, 3-arm, phase II pilot study. Neurooncol Adv. 2021 Dec 27;4(1):vdab188. doi: 10.1093/noajnl/vdab188. eCollection 2022 Jan-Dec. PMID 35156036